CLINICAL TRIAL: NCT02016118
Title: INTRAVESICAL ADMINISTRATION OF COMBINED HYALURONIC ACID (HA) AND CHONDROITIN SULPHATE (CS) vs. STANDARD OF CARE FOR THE TREATMENT OF RECURRENT URINARY TRACT INFECTIONS (RUTIs)
Brief Title: Retrospective Analysis of Ialuril vs. Standard of Care in Recurrent Urinary Tract Infections
Acronym: RAISC-RUTI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Study Group for Urogenital Diseases, Italy (Other)
Responsible Party: Principal Investigator, Massimo Lazzeri, MD, PhD Consultant, Study Group for Urogenital Diseases, Italy
Other Study IDs: RAISC-RUTI
Record Dates: First submitted 2013-10-07; First posted 2013-12-19 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Recurrent Urinary Tract Infections
Keywords: RUTI
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ialuril: Intravesical administration of combined hyaluronic acid (HA) 1.6% and chondroitin sulphate (CS) 2.0% once per week for the first month, followed by one instillation every two weeks for the second month and one instillation per month until stable remission of the symptoms.
  Interventions: Device: Ialuril
- Standard of care: Antimicrobial prophylaxis (continuous or postcoital), as described in the Guidelines on Urological Infections of the European Association of Urology or Immunoactive prophylaxis or Prophylaxis with probiotics or Prophylaxis with cranberry, or combination of these.

INTERVENTIONS:
Device: Ialuril — The treatment is an intravesical administration of combined hyaluronic acid (HA) 1.6% and chondroitin sulphate (CS) 2.0% once per week for the first month, followed by one instillation every two weeks for the second month and one instillation per month until stable remission of the symptoms.
  Groups: Ialuril

SUMMARY:
The purpose of this study is to assess the effectiveness and costs associated with the intravesical administration of combined hyaluronic acid (HA) and chondroitin sulphate (CS) compared to the current standard management of recurrent urinary tract infections in adult women diagnosed with recurrent urinary tract infections (RUTI).

DETAILED DESCRIPTION:
RUTI is defined as at least three episodes of uncomplicated urinary tract infections accompanied by clinical symptoms and documented by urine culture with the isolation of >103 colony forming units (CFU)/ml of an identified pathogen in the last year (M. Grabe, T.E. Bjerklund-Johansen, H. Botto, B. Wullt, M. Çek, K.G. Naber, R.S. Pickard, P. Tenke, F. Wagenlehner. Guidelines on Urological Infections. European Association of Urology 2012).

In order to do so, we will perform a retrospective analysis on prospectively collected patient data in nine European centres.

The treatment schedule for the intravesical administration of combined hyaluronic acid (HA) 1.6% and chondroitin sulphate (CS) 2.0% is one instillation per week for the first month, followed by one instillation every two weeks for the second month and one instillation per month until stable remission of the symptoms.

The current standard management of RUTI in Europe is represented by the antimicrobial prophylaxis (continuous or postcoital), as described in the Guidelines on Urological Infections of the European Association of Urology or Immunoactive prophylaxis or Prophylaxis with probiotics or Prophylaxis with cranberry, or combination of these.

We will collect patient characteristics as age, BMI, sexual activity, employment status, severity of the disease, comorbidities.

Our primary clinical outcome will be the occurrence of objective (bacteriologically confirmed) recurrence within 12 months after the start of the treatment. Other outcomes will be the occurrence of clinical or symptoms based recurrence; the time to objective or symptoms based recurrence, evaluated from the start of the treatment until the first occurrence of an objective or symptoms based urinary tract infection, and the overall number of objective or symptoms based urinary tract infections experienced within 12 months after treatment initiation for RUTI.

Information about health related quality of life at baseline and 12 months will be recorded if available.

In terms of resource utilization, we will record the number of medical visits, number and types of laboratory, imaging and instrumental exams, hospitalization, consumption of pharmaceuticals or instrumental therapies (other than intervention and comparator) used within 12 months since treatment initiation. Number of days absent from work due to RUTI will be recorded when available. Costs will be attributed according to the perspective of the National Healthcare System searching for relevant data sources in each country.

Standard descriptive statistics, such as mean, median, range, and proportions, will be used to summarize patient characteristics and other collected variables. The Chi-Square test will be used to compare differences in proportions and the Mann-Whitney U test to compare continuous variables, with or without logarithmic transformation. The Kaplan-Meier method will be used to estimate time to recurrence outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-75 years old.
* Women diagnosed with recurrent urinary tract infections, defined as at least three episodes of uncomplicated urinary tract infections accompanied by clinical symptoms and documented by urine culture with the isolation of >103 CFU/ml of an identified pathogen in the last year. Uncomplicated or 'simple' UTI is defined as an infection in a person with normal urinary tract and function.

Exclusion criteria:

- Women with complicated urinary tract infections. Complicated urinary tract infection occurs in individuals with functional or structural abnormalities of the genitourinary tract.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will consider women with recurrent urinary tract infections who started their treatments at the Urology Departments at the enrolling centres.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-03 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Urinary tract infection recurrence | within 12 months after treatment initiation
  At least one bacteriologically confirmed urinary tract infection experienced within 12 months after the treatment initiation.

SECONDARY OUTCOMES:
Occurrence of symptomatic urinary tract infection recurrence | within 12 months after treatment initiation
  At least one symptoms based urinary tract infection experienced within 12 months after the treatment initiation.

OTHER OUTCOMES:
Mean direct overall costs | within 12 months after treatment initiation
  Mean overall costs, expressed in euros, comprehensive of costs of each treatment options and other direct medical costs (i.e. visits, additional medical therapies required because of recurrences or adverse events, hospitalization) measured over 12 months after treatment initiation for each cohort of patients.
Number of days absent from work | within 12 months after treatment initiation
  Number of days of absence from work due to the recurrent urinary tract infections within 12 months since the start of the treatment.
Time-to-recurrence | 12 months after treatment initiation
  Time from the start of the treatment until the first occurrence of an objective or symptoms based urinary tract infection

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Lazzeri, PhD, Principal Investigator — Università Vita-Salute San Raffaele
Locations (1):
- Ospedale S. Maria della Misericordia, Perugia, Perugia, Italy

REFERENCES:
- [Background] Naber KG, Bergman B, Bishop MC, Bjerklund-Johansen TE, Botto H, Lobel B, Jinenez Cruz F, Selvaggi FP; Urinary Tract Infection (UTI) Working Group of the Health Care Office (HCO) of the European Association of Urology (EAU). EAU guidelines for the management of urinary and male genital tract infections. Urinary Tract Infection (UTI) Working Group of the Health Care Office (HCO) of the European Association of Urology (EAU). Eur Urol. 2001 Nov;40(5):576-88. doi: 10.1159/000049840. PMID 11752870
- [Derived] Ciani O, Arendsen E, Romancik M, Lunik R, Costantini E, Di Biase M, Morgia G, Fragala E, Roman T, Bernat M, Guazzoni G, Tarricone R, Lazzeri M. Intravesical administration of combined hyaluronic acid (HA) and chondroitin sulfate (CS) for the treatment of female recurrent urinary tract infections: a European multicentre nested case-control study. BMJ Open. 2016 Mar 31;6(3):e009669. doi: 10.1136/bmjopen-2015-009669. PMID 27033958